CLINICAL TRIAL: NCT04448041
Title: A Cluster Randomised Feasibility Study of a Sustainable Nutritional Intervention for Patients Undergoing Cancer Surgery in Low- and Middle-Income Countries
Brief Title: CRANE Feasibility Study: Nutritional Intervention for Patients Undergoing Cancer Surgery in Low- and Middle-Income Countries
Acronym: CRANE
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: CRANE
Record Dates: First submitted 2020-06-11; First posted 2020-06-25 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Malnutrition; Surgery; Cancer
Keywords: Malnutrition; Screening tools; Cancer surgery; Low and middle-income countries (LMIC)
MeSH Terms: conditions — Malnutrition; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Ghana
  Interventions: Other: Malnutrition screening
- India
  Interventions: Other: Malnutrition screening
- Philippines
  Interventions: Other: Malnutrition screening
- Zambia
  Interventions: Other: Malnutrition screening

INTERVENTIONS:
Other: Malnutrition screening — Primary comparison: Prevalence of malnutrition and impact on 30-day outcomes in patients undergoing surgery for cancer

SUMMARY:
Aims: The CRANE feasibility study (A mixed methods study of malnutrition and sustainable nutritional intervention for patients undergoing cancer surgery in low- and middle-income countries) aims to investigate the identification of pre-operative malnourishment, data collection methods and acceptability of a nutritional intervention for a future trial to improve outcomes after cancer surgery in low- and middle-income countries (LMICs).

1. To identify and validate the most relevant nutritional screening tool for patients in LMICs undergoing surgery for cancer;
2. To identify a low cost sustainable nutritional intervention for patients in LMICs undergoing surgery for cancer;
3. To establish the feasibility of delivering a randomised trial of a sustainable nutritional intervention for patients in LMICs undergoing surgery for cancer.

Design: A mixed-methods study comprising of qualitative work including focus groups and interviews, trial of data collection and validation to test feasibility in clinical practice

Participants: Patients undergoing elective surgery for suspected cancer in LMICs

Outcomes Work package (WP) 1: The primary deliverable is the identification of a relevant, pragmatic, and acceptable nutritional screening tool.

WP 2: The primary deliverable is the identification of a low-cost and sustainable nutritional intervention. Focus groups and interviews will be held with patients and clinicians to explore the sustainability, implementation and acceptability of screening and interventions.

WP 3: The primary outcome will be to determine feasibility and acceptability of trial design. A number of outcome assessments and data collection instruments will be evaluated for feasibility, including anthropometric parameters and patient outcomes (30-day mortality, major post-operative complications, length of hospital stay and quality of life). A final study design, analysis plan, and health economic plan will be developed.

Sample size: For this feasibility study, the investigators will conduct multidisciplinary focus groups and interviews, perform and validate malnutrition screening in 200 patients across four countries and record patient 30-day outcomes. This will also include the time taken to collect data on 200 eligible patients. This sample size has been informed from previous malnutrition data originating from a large prospective international multicentre observational cancer study (GlobalSurg 3).

ELIGIBILITY:
Inclusion Criteria:

* Hospitals in LMICs who undertake planned (elective) cancer surgery for cancer.
* Patients over 18 years of age (or the age of majority for the country);
* Patients undergoing planned (elective) surgery for cancer;
* Patients undergoing surgery where the intent is either curative or palliative;
* Patients must be able and willing to provide written informed consent (signature or a fingerprint).

Exclusion Criteria:

* Children (below age of majority for the country);
* Patients undergoing emergency surgery;
* Any operative indication other than cancer;
* Patients unable to provide written informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for cancer in four partner LMIC countries are eligible
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of malnutrition | Immediately prior to surgery
  Malnutrition as measured using validated screening tools
30-day mortality rate | 30 days from surgery
  Death within 30 days of surgical procedure

SECONDARY OUTCOMES:
30-day complication rate | 30 days from surgery
  Defined with by Clavien-Dindo grade III or IV
Length of stay | 30 days from surgery
  Length of hospital admission
Re-operation rate | 30 days from surgery
  Re-operation within 30 days of surgical procedure
Quality of life following surgery (EQ-5D-5L / WHODAS questionnaire (36 item)) | 30 days from surgery
  Short-term quality of life for patients following surgery
Readmission rates | 30 days from surgery
  Readmission within 30 days of surgery
Recruitment rate | Through study duration, up to one year
  Time taken to recruit 200 patients

CONTACTS AND LOCATIONS:
Overall Officials: Ewen Harrison, Principal Investigator — University of Edinburgh
Locations (11):
- Ghana (2):
  - Cape Coast Teaching Hospital, Cape Coast
  - Tamale Teaching Hospital, Tamale
- India (5):
  - Tata medical Centre, Kolkata
  - CMC Ludhiana, Ludhiana
  - Padhar Hospital, Pādhar
  - AIIMS, Rishikesh
  - Christian Medical College, Vellore
- Philippines (4):
  - Medical Center, Manila
  - Philippine General Hospital (UP-PGH), Manila
  - Rizal Medical Center, Manila
  - The Medical City Hospital, Manila

IPD SHARING:
Plan to Share IPD: Yes
Derived anonymised data at the patient-level may be able to be made available for sharing
Supporting Information: Study Protocol, SAP, Analytic Code